NCT NUMBER: DATE:28.11.25

## **RESULTS FORM**

TITLE/PURPOSE OF THE STUDY: EVALUATE THE EFFICACY OF SUBGINGIVAL APPLICATION OF 1.2% LOVASTATIN GEL AS AN ADJUNCT TO CONVENTIONAL NON-SURGICAL PERIODONTITIS THERAPY IN GENERALLY HEALTHY NON-SMOKING AND SMOKING PATIENTS FROM CENTRAL EUROPE: A RANDOMIZED SPLIT-MOUTH CONTROL TRIAL

Intra-group comparsion of the measurments of clinical parameters (mean  $\pm$  SD) at the baseline and 3 and 6 months later (in mm)

| Parameters | Group 1 (non-smokers) | | Group 2 (smokers) | |
|---|---|---|---|---|
| | Placebo | Lovastatin | Placebo | Lovastatin |
| PPD | | <u> </u> | | |
| Baseline | | | | |
| 3 months | | | | |
| 6 months | | | | |
| CAL | | | | |
| Baseline | | | | |
| 3 months | | | | |
| 6 months | | | | |

Intra-group comarsion of the measurments of radiographic parameters (mean  $\pm$  SD) at the baseline and 6 months later (in mm)

| Parameter | Group 1 (non-smokers) | | Group 2 (smokers) | |
|---|---|---|---|---|
| | Placebo | Lovastatin | Placebo | Lovastatin |
| IBD | | | | |
| Baseline | | | | |
| 3 months | | | | |
| 6 months | | | | |